CLINICAL TRIAL: NCT02587494
Title: Role of Early Cardiac Catheterization in Cardiac Arrest
Brief Title: Cardiac Catheterization in Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106834
Record Dates: First submitted 2015-08-27; First posted 2015-10-27 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Cardiac Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cardiac catheterization (Active Comparator): Cardiac catheterization performed as early as possible, within 12h post ROSC following OHCA, with possible PCI during mild therapeutic hypothermia or apyrexia
  Interventions: Procedure: Cardiac catheterization
- Medical arm (No Intervention): Initial therapy does not include cardiac catheterization. Cardiac catheterization with possible PCI is allowed after completion of mild therapeutic hypothermia or apyrexia for >24h post ROSC.

INTERVENTIONS:
Procedure: Cardiac catheterization — Cardiac catheterization / coronary angiography is a diagnostic procedure used to define the coronary anatomy and presence of obstructive coronary lesions or culprit lesions. According to the findings, it may lead to percutaneous coronary intervention (PCI) using stents
  Other Names: Coronary angiography
  Arms: Early cardiac catheterization

SUMMARY:
This is a pilot study that will lead to a large randomized control trial (RCT), to assess whether early versus late or no cardiac catheterization is associated with improved outcomes in out-of-hospital cardiac arrest (OHCA) patients.

DETAILED DESCRIPTION:
A pilot multicenter RCT.

The objectives of the study are:

To assess whether early (within 12 hours) cardiac catheterization is associated with improved survival, neurologic and cardiovascular outcomes in OHCA patients.

Patients will be randomized 1:1 to early cardiac catheterization, performed as early as possible, within 12h post return of spontaneous circulation (ROSC) following OHCA, or to standard practice, which may include medical management without cardiac catheterization or late cardiac catheterization after completion of therapeutic hypothermia. Percutaneous coronary intervention (PCI) is recommended for culprit lesions found on diagnostic angiography. All patients will undergo therapeutic hypothermia started as soon as possible with target temperature below 36°C according to local practice. Other medical management will be according to standard of care

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale score <8 on hospital admission following OHCA of presumed cardiac cause.
* Initial rhythm ventricular tachycardia (VT) / ventricular fibrillation (VF), who achieved ROSC sustained for >20 consecutive minutes

Exclusion Criteria:

* ST-elevation on any of the ECGs post resuscitation
* Hypothermia <30°C
* Interval from ROSC to screening of >12h
* Suspected or known acute intracranial hemorrhage or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite of death and poor neurologic outcomes ( Cerebral Performance Category [CPC] score 3-5). | 30 days

SECONDARY OUTCOMES:
Death | 30 day
CPC score | up to 30 days
Acute kidney injury- creatinine levels | 48 hours
  Number of participants with increase in serum creatinine of ≥44.2 μmol/L, or a 25% relative rise in creatinine, within 48 h after contrast exposure42
Myocardial infarction - according to cardiac troponin levels | 30 days
  Number of participants with myocardial infarction post percutaneous coronary interventions, in accordance with the universal definition of myocardial infarction.
Stent thrombosis by pathology or angiography | 30 days
  Number of participants with definite stent thrombosis confirmed by angiography or pathology according to the Academic research consortium criteria
Bleeding - according to Hb levels | 30 days
  Number of participant with overt bleeding according to Academic Research Consortium criteria
Composite of death and poor neurologic outcome | 1 year
Stroke - imaging or pathology | 30 days
  New stroke following hypothermia confirmed by imaging (computer tomography or magnetic resonance imaging)
Heart failure (NYHA 3-4) | 30 days
Estimated cost per patient according to length of stay and procedures performed | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada